CLINICAL TRIAL: NCT07221487
Title: Low Versus Standard Intra-Abdominal Pressure During Gynecologic Laparoscopy: A Randomized Controlled Trial of Postoperative Pain and Recovery Outcomes
Brief Title: Comparing Intra-Abdominal Pressure During Gynecologic Laparoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nassau University Medical Center (Other)
Responsible Party: Principal Investigator, PETR ITZHAK, Attending Physician, Nassau University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-300
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Gynecologic Surgical Procedures
Keywords: pain; abdominal pressure
MeSH Terms: conditions — Pain | interventions — Lower Body Negative Pressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard-pressure group (Active Comparator): 15 mmHg pressure
  Interventions: Procedure: abdominal pressure
- low-pressure group (Experimental): 8 mmHg
  Interventions: Procedure: abdominal pressure

INTERVENTIONS:
Procedure: abdominal pressure — type of intra-abdominal pressure of either standard or low pressure

SUMMARY:
The goal of this clinical trial is to learn if the level of intra-abdominal pressure during benign gynecologic laparoscopic surgery impacts postoperative pain.

The main question it aims to answer is:

• Does use of low (8 mmHg) versus standard (15 mmHg) intra-abdominal pressure impact postoperative pain?

Researchers will compare the use of low (8 mmHg) versus standard (15 mmHg) intra-abdominal pressure.

Participants will:

* Undergo their regular scheduled gynecologic laparoscopic surgery
* Complete pain measures one hour, 3 hours, and 24 hours after surgery

DETAILED DESCRIPTION:
Participants will be randomized into one of two experimental groups using a computer-generated allocation list: a low-pressure group (8 mmHg) or a standard-pressure group (15 mmHg). As part of standard care, many surgeons more often use 15 mmHg which is why this is named as our standard-pressure group. Some surgeons use low-pressure varying from 8 mmHg through 12 mmHg which is why our 8 mmHg is named the low-pressure group. The 8 mmHg is the most common acceptable low-pressure approach reported in the surgical literature. All surgeries will begin with standard insufflation at 15 mmHg to achieve safe abdominal access. Once the operative field is established, if necessary, the pressure will be adjusted according to the assigned group. For those surgeons who use 8 mmHg, standard care is to start at 15 mmHg and then to adjust to the lower pressure of 8 mmHg. Our proposed approach is consistent with standard clinical protocol. General anesthesia will be administered per institutional protocol, and local anesthetic will be applied to all trocar sites.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing benign gynecologic laparoscopic surgery with eligible procedures, including the following.
* Salpingectomy
* Cystectomy
* Oophorectomy
* Myomectomy
* Hysterectomy.
* Only those who speak English or Spanish will be recruited, as our validated questionnaires are only available in those languages.

Exclusion Criteria:

* Participants with the following diseases will be excluded due to their diseases having pain that may strongly interfere with their perception of pain in the area of surgery.
* Arthritis
* Gout
* Metastatic cancer
* Pelvic floor disease
* Headache disorders
* Herpes zoster or shingles
* Frozen shoulder
* Complex regional pain syndrome (CRPS)
* Slipped disc
* Sickle cell disease
* Sciatica
* Trigeminal neuralgia
* Fibromyalgia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
PAIN OUT questionnaire | Perioperative/Periprocedural: Three hours after surgery completed
  Self-report questionnaire to patient participants focusing on shoulder pain with a total composite score from 12 items. Minimum score is 0 and maximum score is 120. Higher scores indicate greater pain levels.

SECONDARY OUTCOMES:
PAIN OUT questionnaire | Perioperative/Periprocedural: 24 hours after surgery completed
  Self-report questionnaire to patient participants focusing on shoulder pain with a total composite score from 12 items. Minimum score is 0 and maximum score is 120. Higher scores indicate greater pain levels.
Numerical rating scale for pain location in the abdomen | Perioperative/Periprocedural: One hour after surgery
  One item to patient participants to rate the abdominal pain from 0 (no pain) to 10 (worst pain)
Numerical rating scale for pain location in the shoulder | Perioperative/Periprocedural: One hour after surgery
  One item to patient participants to rate the shoulder pain from 0 (no pain) to 10 (worst pain)
Visual analog scale for pain location in the abdomen | Perioperative/Periprocedural: Three hours after surgery completed
  One item to patient participants to rate the abdominal pain from 0 (no pain) to 10 (worst pain)
Visual analog scale for pain location in the abdomen | Perioperative/Periprocedural: 24 hours after surgery completed
  One item to patient participants to rate the abdominal pain from 0 (no pain) to 10 (worst pain)
Length of hospital stay | Perioperative/Periprocedural
  Length of hospital stay for the patient participants after surgery completed measured in minutes. Longer stay defined as greater number of minutes
Complications | Perioperative/Periprocedural
  Presence of nausea or vomiting after surgery in patient participants. Yes responses indicate the presence of complications
Hospital Readmission | Perioperative/Periprocedural
  Hospital readmission to patient participants within 30 days after surgery completed. Yes indicates a hospital readmission
Use of non-medicine methods to relieve pain | Perioperative/Periprocedural
  Provided a checklist to patient participants of non-medicine choices such as cold pack, meditation, prayer, massage, distraction like watching television. A yes to any of these choices indicates use of non-medicine methods to relieve pain
Overall Quality of Surgical Visual Field | Perioperative/Periprocedural
  Question to the surgeon with choices rating the overall surgical conditions throughout the procedure from extremely poor with a choice of 1 to optimal with a choice of 5. Higher scores indicate a better overall quality of surgical visual field

CONTACTS AND LOCATIONS:
Overall Officials: Petr Itzhak, DO, Principal Investigator — Nassau University Medical Center
Locations (1):
- Nassau University Medical Center, East Meadow, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentfied data based upon a reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study using data is published
Access Criteria: Academic researchers

REFERENCES:
- [Background] Reijnders-Boerboom GTJA, Albers KI, Jacobs LMC, Helden EV, Rosman C, Diaz-Cambronero O, Mazzinari G, Scheffer GJ, Keijzer C, Warle MC. Low intra-abdominal pressure in laparoscopic surgery: a systematic review and meta-analysis. Int J Surg. 2023 May 1;109(5):1400-1411. doi: 10.1097/JS9.0000000000000289. PMID 37026807